CLINICAL TRIAL: NCT03635385
Title: Comparison of ANCA and Anti-GBM Auto-antibodies Removal Kinetics Between Plasma Exchanges and Immunoadsorption in Patients With ANCA-associated Vasculitis or Anti-GBM Disease
Acronym: CINEVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-31; 2018-A00510-55 (Other: Ansm)
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma exchange (PE) technic patient group (Active Comparator)
  Interventions: Procedure: Apheresis technics
- Immunoadsorption technic patient group (Active Comparator)
  Interventions: Procedure: Apheresis technics

INTERVENTIONS:
Procedure: Apheresis technics — Blood draw will be performed for anti bodies dosages

SUMMARY:
Anti-neutrophil cytoplasmic antibodies (ANCA), directed against myeloperoxidase (MPO) and against proteinase 3 (PR3), have a pathogenic role during ANCA (AAV) vasculitis. Glomerular basement membrane (MBG) antibodies also have a direct pathogenic role in Goodpasture's syndrome and anti-MBG antibody glomerulonephritis (GN). In some patients, the severity of renal and / or pulmonary involvement justifies the rapid purification of these autoantibodies by an apheresis procedure, while waiting for the effect of immunosuppressive treatments aimed at reducing their production. During vasculitis, plasma exchange (PE) is recommended in patients with severe renal impairment or intra-alveolar hemorrhage (2012 KDIGO Clinical Practice Guideline for Glomerulonephritis).

Given certain disadvantages related to plasma exchanges (low volume of purified plasma, non-selective technique for immunoglobulins (Ig), need for replacement solute, induction of coagulation disorders), immunoadsorption (IA), already used in transplantation, has been developed in these indications. IA has indeed greater selectivity for Ig with a probable better purification capacity due to higher volumes of plasma treated per session. The price of IA is however higher than that of EP.

These two apheresis techniques, EP and IA, are commonly used in France during severe forms of vasculitis ANCA or anti-MBG, without the superiority of one or the other has been demonstrated. As a result of higher plasma volumes being purified, AI may allow faster purification of pathogenic antibodies. No studies to date have specifically compared the purification kinetics of these antibodies between EP and IA.

The CINEVAS study (VAScularite Antibody Purification CINetic) is a multicentric pilot study whose main objective is to compare the purification kinetics of ANCA (anti-MPO or anti-PR3) and / or anti- MBG in patients treated with EP versus those treated with IA

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with ANCA vasculitis with positive anti-MPO or anti-PR3 antibodies, or patient with Goodpasture syndrome or anti-MBG antibody glomerulonephritis
* Patient for whom the investigating physician retains the indication of apheresis
* Induction treatment with corticosteroids and cyclophosphamide or rituximab

Exclusion Criteria:

* Pregnancy or breastfeeding
* Vasculitis without anti-MPO, anti-PR3 or anti-MBG
* Severe anemia (hemoglobin <7 g / dL) contraindicates additional blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Percent of Anti-glomerular basement membrane anitibodies | 12 months
  Comparison of anti-glomerular basement membrane anitibodies dosage between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assisatance Publique Hôpitaux de Marseille, Marseille, France